CLINICAL TRIAL: NCT03957928
Title: Effects of Fresh Mango Pulp Consumption on Satiety and Cardiometabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HS-2019-0034
Record Dates: First submitted 2019-04-25; First posted 2019-05-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Satiety
MeSH Terms: interventions — Mangifera indica extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low fat cookies (Active Comparator): Subjects consume 100 kcal of low fat cookies daily for 12 weeks.
  Interventions: Other: Low fat cookie
- Mango fruit (Experimental): Subjects consume 100 kcal of mango fruit daily for 12 weeks.
  Interventions: Other: Mango fruit

INTERVENTIONS:
Other: Low fat cookie — to determine the effects of low fat cookie consumption on satiety and metabolic parameters in overweight/obese adults
  Arms: Low fat cookies
Other: Mango fruit — to determine the effects of fresh mango pulp consumption on satiety and metabolic parameters in overweight/obese adults
  Arms: Mango fruit

SUMMARY:
The objective of the study is to determine the effects of fresh mango pulp consumption on satiety and metabolic parameters in overweight/obese adults.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old
* BMI 27-40

Exclusion Criteria:

* Smoker
* Pregnant woman
* Required dietary supplement use
* Required medication of metabolic disorders
* Allergy to mango or gluten

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change of satiety | 0, 20, 40, 60, 90 and 120 minutes post snack consumption
  Change of hunger feeling (appetite) will be examined using visual analog scale (0-10): 0 least and 10 greatest
Change of glucose level | 0, 30, 60, 90 and 120 minutes post snack consumption; baseline and week 12
  Change of blood glucose response will be determined to examine effects of mango consumption vs low fat cookie consumption
Change of insulin level | 0 and 60 minutes post snack consumption, baseline and week 12
  Change of blood insulin level will be determined to examine effects of mango consumption vs low fat cookie consumption

SECONDARY OUTCOMES:
Change of microbiome | Baseline, week 4 and week12
  Change of microbiome diversity will be determined to examine effects of mango consumption vs low fat cookie consumption

CONTACTS AND LOCATIONS:
Locations (1):
- School of Exercise and Nutritional Sciences, SDSU, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosas M Jr, Pinneo S, O'Mealy C, Tsang M, Liu C, Kern M, Hooshmand S, Hong MY. Effects of fresh mango consumption on cardiometabolic risk factors in overweight and obese adults. Nutr Metab Cardiovasc Dis. 2022 Feb;32(2):494-503. doi: 10.1016/j.numecd.2021.11.001. Epub 2021 Nov 12. PMID 34953634
- [Derived] Pinneo S, O'Mealy C, Rosas M Jr, Tsang M, Liu C, Kern M, Hooshmand S, Hong MY. Fresh Mango Consumption Promotes Greater Satiety and Improves Postprandial Glucose and Insulin Responses in Healthy Overweight and Obese Adults. J Med Food. 2022 Apr;25(4):381-388. doi: 10.1089/jmf.2021.0063. Epub 2021 Nov 23. PMID 34813369